CLINICAL TRIAL: NCT02293265
Title: Identification and Description of Severe Asthma Patients in a Cross-sectional Study-the IDEAL Study
Brief Title: Cross-sectional Study for Identification and Description of Severe Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 201722
Record Dates: First submitted 2014-10-27; First posted 2014-11-18 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: mepolizumab; omalizumab; SB-240563; Severe Asthma; reslizumab
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-drug interventional group (Other): All enrolled participants will provide a blood sample, spirometry , and feedback on their severe asthma symptoms via questionnaires, and health related quality of life and burden of illness through response to self-administered questionnaires. No investigational product will be administered to participants.
  Interventions: Drug: Short Acting Beta Agonist (SABA)

INTERVENTIONS:
Drug: Short Acting Beta Agonist (SABA) — Participants requiring a spirometry measurement will be administered a SABA in a metered dose inhaler (MDI) during the reversibility assessments

SUMMARY:
This will be a non-drug interventional cross-sectional study, where the screening visit and study visit can occur on the same day. Investigational product will not be administered. Approximately 790 subjects with severe asthma will be screened to achieve a total of at least 750 evaluable study subjects. The study will not include a run-in or follow-up period. This study will provide a more reliable description of the severe asthma patient landscape with respect to the potential eligibility for treatment with mepolizumab, omalizumab, and reslizumab. This study aims to estimate the potential overlap of patients eligible for treatment with mepolizumab and those eligible for treatment with omalizumab and/or reslizumab. Additionally, the current study will also ascertain and describe reslizumab eligibility with respect to both mepolizumab and omalizumab, in the severe asthma patient population.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age at study visit.
* Participants eligible for enrolment and entry into the study must meet the following definition of severe asthma, which is based on the definition of severe asthma described in the European Respiratory Society/ American Thoracic Society (ERS/ATS) Guidelines for severe asthma: Asthma which requires treatment with guideline suggested medications for Global Initiative for Asthma (GINA) steps 4-5 asthma for the previous year (i.e., at least 12 months).

Patients must be treated with high dose ICS PLUS at least one of the following: LABA, leukotriene modifier, theophylline, or continuous or near continuous systemic corticosteroid (i.e., maintenance systemic corticosteroid for ≥50% of the previous year).

SPECIAL CIRCUMSTANCE: If patient is on a fixed dose combination medication, then the maximum recommended dose of the ICS/LABA combination per local label is acceptable.

* Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Participants must be able to read, comprehend, and write at a level sufficient to complete study related materials. A parent or legal guardian must provide informed consent for participants less than 18 years of age at study visit (or less than minimum age to be considered an adult per local laws).

Exclusion Criteria:

Participants who have participated in an interventional clinical trial for asthma within the past 12 months prior to Visit 1 (NOTE: subjects participating in an observational study where an investigational product or procedure is not administered will not be subject to this exclusion criteria)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of severe asthma patients eligible for one or more biologic treatments for asthma | Day 1
  Biologic treatments for asthma will include mepolizumab (anti-Interleukin [IL] 5), omalizumab (anti-immunoglobulin E [IgE]), and reslizumab (anti-IL5).

SECONDARY OUTCOMES:
Mean and median frequency of planned and unplanned asthma-related healthcare resource utilization in the prior 12 months | Day 1
Mean and median Charlson Comorbidity Index score | Day 1
  The Charlson Comorbidity Index is a score that is based on age and the presence of 19 comorbidities. The mean and median Charlson Comorbidity Index score will be calculated and reported
Mean pre-bronchodilator forced expiratory volume in 1 sec (FEV1)/forced vital capacity (FVC) ratio | Day 1
  Spirometry assessment will be performed with mean pre- and post-bronchodilator FEV1/FVC, pre- and post-bronchodilator FEV1 and FVC, and airway reversibility
Mean post-bronchodilator FEV1/FVC ratio | Day 1
  Spirometry assessment will be performed with mean pre- and post-bronchodilator FEV1/FVC, pre- and post-bronchodilator FEV1 and FVC, and airway reversibility
Mean pre-bronchodilator FEV1 | Day 1
  Spirometry assessment will be performed with mean pre- and post-bronchodilator FEV1/FVC, pre- and post-bronchodilator FEV1 and FVC, and airway reversibility
Mean post-bronchodilator FEV1 | Day 1
  Spirometry assessment will be performed with mean pre- and post-bronchodilator FEV1/FVC, pre- and post-bronchodilator FEV1 and FVC, and airway reversibility
Mean pre-bronchodilator FVC | Day 1
  Spirometry assessment will be performed with mean pre- and post-bronchodilator FEV1/FVC, pre- and post-bronchodilator FEV1 and FVC, and airway reversibility
Mean post-bronchodilator FVC | Day 1
  Spirometry assessment will be performed with mean pre- and post-bronchodilator FEV1/FVC, pre- and post-bronchodilator FEV1 and FVC, and airway reversibility
Mean and median levels of blood eosinophils | Day 1
Mean and median levels of total IgE | Day 1
Mean and median levels of specific IgE | Day 1
Descriptive statistics for asthma Control Questionnaire (ACQ-5) | Day 1
Descriptive statistics for St. George's Respiratory Questionnaire (SGRQ) | Day 1
Descriptive statistics for Asthma Quality of Life Questionnaire (AQLQ-S) | Day 1
Descriptive statistics for EuroQol 5D (EQ-5D-5L) | Day 1
Descriptive statistics for Work Productivity and Activity Impairment Index: General Health (WPAI-GH) | Day 1
Descriptive statistics for Asthma Symptom Utility Index (ASUI) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (65):
- United States (21):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Corning, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
- GSK Investigational Site, Coffs Harbour, New South Wales, Australia
- Canada (12):
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Grimsby, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, St-Charles-Borromée, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- France (14):
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Tarbes
  - GSK Investigational Site, Villefranche-sur-Saône
- Germany (8):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- United Kingdom (9):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Crawley
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Radstock, Bath
  - GSK Investigational Site, Salford
  - GSK Investigational Site, Trowbridge

REFERENCES:
- [Derived] Mullerova H, Cockle SM, Gunsoy NB, Nelsen LM, Albers FC. Clinical characteristics and burden of illness among adolescent and adult patients with severe asthma by asthma control: the IDEAL study. J Asthma. 2021 Apr;58(4):459-470. doi: 10.1080/02770903.2019.1708095. Epub 2020 Jan 9. PMID 31874051
- [Derived] Nelsen LM, Cockle SM, Gunsoy NB, Jones P, Albers FC, Bradford ES, Mullerova H. Impact of exacerbations on St George's Respiratory Questionnaire score in patients with severe asthma: post hoc analyses of two clinical trials and an observational study. J Asthma. 2020 Sep;57(9):1006-1016. doi: 10.1080/02770903.2019.1630640. Epub 2019 Jun 28. PMID 31251094
- [Derived] Albers FC, Mullerova H, Gunsoy NB, Shin JY, Nelsen LM, Bradford ES, Cockle SM, Suruki RY. Biologic treatment eligibility for real-world patients with severe asthma: The IDEAL study. J Asthma. 2018 Feb;55(2):152-160. doi: 10.1080/02770903.2017.1322611. Epub 2017 Jun 16. PMID 28622052